CLINICAL TRIAL: NCT05744999
Title: THE COCONUT TECHNIQUE - A NEW METHOD TO PERFORM SAFE CHOLECYSTECTOMY FOR ACUTE CHOLECYSTITIS: Our Initial Experience
Brief Title: HOW TO PERFORM SAFELY CHOLECYSTECTOMY FOR ACUTE CHOLECYSTITIS
Status: Completed | Type: Observational
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Isidoro Di Carlo, MD, PhD, FACS, Professor, University of Catania
Other Study IDs: IDC-002
Record Dates: First submitted 2023-02-15; First posted 2023-02-27 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Cholecystectomy
Keywords: acute cholecystitis; cholecystectomy; cystic duct
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with the reported technique: Two females and 1 male with a mean age of 50 years were diagnosed by CT scan with stage II acute cholecystitis according to the Tokyo guidelines and were operated on within three days of symptom onset
  Interventions: Procedure: Coconut technique

INTERVENTIONS:
Procedure: Coconut technique — We recently developed a simple but effective laparoscopic technique to approach and ligate the cystic duct in cases of difficult acute cholecystitis. Three to four centimeters of the inflamed gallbladder wall was then cut using an electrocautery hook. An incision was made in a safe zone at the junction of the infundibulum and the body of the gallbladder. The separation between the outer layer and inner layer was searched. This clear identification of the confluence between the cystic duct and the body of the gallbladder represents the way to determine if the procedure was safely completed using the current technique. After successful identification, the cystic duct was clipped. The gallbladder can then be lifted and turned over, leaving the unidentified CBD untouched, and cholecystectomy can be carefully performed as usual. The inflamed posterior wall remained attached to the gallbladder bed of the liver.

SUMMARY:
The aim of this manuscript is to illustrate a new method permitting safe cholecystectomy in terms of complications with respect to the common bile duct (CBD).

The core of this new technique is identification of the continuity of the cystic duct with the infundibulum. The cystic duct can be identified between the inner gallbladder wall and inflamed outer wall.

In the last 2 years, 3 patients have been treated with the reported technique without complications.

Among the various cholecystectomy procedures, this is a new approach that ensures the safety of the structures of Calot's triangle while providing the advantages gained from total removal of the gallbladder.

ELIGIBILITY:
Inclusion Criteria:

* stage II acute cholecystitis according to the Tokyo guidelines
* symptom onset

Exclusion Criteria:

- stage I cholecystectomy

Max Age: 50 Years | Sex: All
Age Groups: Child, Adult
Study Population: Two females and 1 male with a mean age of 50 years were diagnosed by CT scan with stage II acute cholecystitis according to the Tokyo guidelines and were operated on within three days of symptom onset.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
A new technique of subtotal cholecystectomy | two years
  Three to four centimeters of the inflamed gallbladder wall was then cut using an electrocautery hook. An incision was made in a safe zone at the junction of the infundibulum and the body of the gallbladder. The separation between the outer layer and inner layer was searched. This clear identification of the confluence between the cystic duct and the body of the gallbladder represents the way to determine if the procedure was safely completed using the current technique. After successful identification, the cystic duct was clipped.

CONTACTS AND LOCATIONS:
Locations (1):
- Isidoro Di carlo, Catania, CT, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT05744999/Prot_000.pdf